CLINICAL TRIAL: NCT02219464
Title: Nasopharyngeal Versus Nasal Cannula Oxygen Supplementation in Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Bret Alvis, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130627
Record Dates: First submitted 2014-08-12; First posted 2014-08-19 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2016-05

CONDITIONS: Oxygen Administration During Deep Sedation
Keywords: nasopharyngeal catheter; nasal cannula
MeSH Terms: interventions — Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasopharyngeal catheter (Active Comparator): Patients in this arm will receive oxygen supplementation through the use of a Nasopharyngeal catheter. Sedation will be standardized to ensure consistency between groups.
  Interventions: Device: Nasopharyngeal catheter; Procedure: Oxygen Supplementation; Procedure: Sedation
- Nasal Cannula (Other): Patients will receive oxygen supplementation through the use of a traditional nasal cannula. Sedation will be standardized to ensure consistency between groups.
  Interventions: Device: Nasal Cannula; Procedure: Oxygen Supplementation; Procedure: Sedation

INTERVENTIONS:
Device: Nasopharyngeal catheter
  Arms: Nasopharyngeal catheter
Device: Nasal Cannula
  Arms: Nasal Cannula
Procedure: Oxygen Supplementation — Initially set at 3 liters/minute
Procedure: Sedation — Midazolam 2mg IV, Fentanyl 100mcg IV, Propofol 100 mcg/kg/min. Additional doses of propofol at the discretion of the attending anesthesiologist.

SUMMARY:
The investigators plan to conduct a randomized, controlled trial comparing nasopharyngeal oxygen supplementation to traditional nasal cannula in patients undergoing oral surgery under moderate sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 16 years of age
* Patients who present for oral surgery or esophagoduodenography and colonoscopy
* Patients who undergo intravenous sedation

Exclusion Criteria:

* Patients who require endotracheal intubation
* ASA class 4 or higher
* Existing esophageal disease such as a perforation or varices

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Alvis, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nasopharyngeal Catheter: Patients in this arm will receive oxygen supplementation through the use of a Nasopharyngeal catheter. Sedation will be standardized to ensure consistency between groups.
  Nasopharyngeal catheter
  Oxygen Supplementation: Initially set at 4 liters/minute
  Sedation: Propofol infusion at 100mcg/kg/min and any increase in propofol was at the discretion of the attending anesthesiologist.
- Nasal Cannula: Patients will receive oxygen supplementation through the use of a traditional nasal cannula. Sedation will be standardized to ensure consistency between groups.
  Nasal Cannula
  Oxygen Supplementation: Initially set at 4 liters/minute
  Sedation: Propofol infusion at 100mcg/kg/min and any increase in propofol was at the discretion of the attending anesthesiologist.
Period: Overall Study
Arm/Group | Nasopharyngeal Catheter | Nasal Cannula
Started | 30 | 30
Completed | 27 | 30
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — case cancelled | 1 | 0
Not completed — catheter malfunction | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasopharyngeal Catheter | Nasal Cannula | Total
Number analyzed (Participants) | 27 | 30 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 8 | 10 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 15 | 16 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27 | 30 | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Oxygen Saturations Below 92%
Time Frame: During surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Nasopharyngeal Catheter | Nasal Cannula
Number analyzed (Participants) | 27 | 30
Participants | 3 | 12

2. Secondary Outcome: Number of Participants Who Needed Airway Assistance Interventions
Description: (jaw lift, tongue retraction, oral airway placement, mask ventilation, increase in oxygen flow rate, ect.).
Time Frame: During surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Nasopharyngeal Catheter | Nasal Cannula
Number analyzed (Participants) | 27 | 30
Participants | 4 | 17

ADVERSE EVENTS:
Time Frame: Adverse events were monitoring for the entire procedure all the way through the patients discharge from the post-anesthesia care unit. This would average around 4 hours of time; however, no time limit was placed on our adverse event monitoring. Once the procedure started to the point they were taken to their form of transportation, each subject was monitored for an adverse event.
Description: The data collection individual would report to the primary investigator and submit report to the Vanderbilt University Institution Review Board.
Arm/Group | Nasopharyngeal Catheter | Nasal Cannula
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/30
Other Adverse Events (participants affected / at risk) | 1/26 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasopharyngeal Catheter (N=26) | Nasal Cannula (N=30)
Nose Bleed (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Nose Bleed from NasoPharyngeal Catheter Placement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes